CLINICAL TRIAL: NCT05058898
Title: A One Health Study of Monkeypox Human Infection, Animal Reservoir, Disease Ecology and Diagnostic Tools
Brief Title: A One Health Study of Monkeypox Human Infection
Acronym: AFRIPOX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de Bangui (Ambiguous)
Responsible Party: Sponsor
Other Study IDs: 2019-047
Record Dates: First submitted 2021-09-24; First posted 2021-09-28 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Monkeypox Virus Infection
Keywords: epidemiology; outbreak investigation; anthropology,; animal reservoir; zoonotic disease; field diagnosis
MeSH Terms: conditions — Mpox, Monkeypox; Zoonoses | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, scabs and pus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Risk factors transmission cases: Human cases of monkeypox confirmed by PCR
  Interventions: Other: blood samples; Other: Scabs and pus samples
- Risk factors transmission contacts and co-exposures: Human contact of confirmed monkeypox cases
  Interventions: Other: blood samples
- Serological follow up cases: Human cases of monkeypox confirmed by PCR from Lobaye region
  Interventions: Other: blood samples; Other: Scabs and pus samples
- Serological follow up contacts and co-exposures: Human contact of confirmed monkeypox cases from Lobaye region adjusted for age, month of the year and village of origin
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — 5 mL
Other: Scabs and pus samples — if available
  Groups: Risk factors transmission cases; Serological follow up cases

SUMMARY:
This multidisciplinary project aim to understand the epidemiology of the monkeypox in Central African Republic through the identification of the animal reservoir, the clinical and epidemiological description of the human outbreak, through an ethnological approach around risk factors of the disease and through an ecological approach of the ecological context of emergence, and the improvement of biological diagnosis.

DETAILED DESCRIPTION:
This project is composed by monkyepox disease outbreak investigation in the CAR following national surveillance framework.

ELIGIBILITY:
Inclusion Criteria:

* Human population in villages affected by monkeypox epidemics: patients who developed monkeypox and their contacts
* Health care personnel (paramedics, nurses, doctors) who work or have worked in affected villages
* Traditional healers, diviners
* Members of villages affected by past monkeypox epidemics

Exclusion Criteria:

* area not accessible to investigation
* refusal to participate
* inability to obtain consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The populations concerned by the study correspond to the sedentary populations known as "Bantus" and the more mobile populations known as "pygmies. These populations belong to different ethno-linguistic groups with more or less specific forest uses and subsistence practices: some are slash-and-burn farmers (Ngbaka, Bagando, Monzombo), others are more mobile and traditionally hunter-gatherers, but now practice agriculture (Bayaka "Pygmies").
  Translated with www.DeepL.com/Translator (free version)
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of monkeypox cases occuring following interhuman exposures | 36 months
  through a quantitative case-control study with an odds ratio of >3 for an exposure factor for human-to-human transmission.
Proportion of monkeypox cases occuring following zoonotic exposures | 36 months
  through a quantitative case-control study with an odds ratio of >3 for an exposure factor for zoonotic transmission.

SECONDARY OUTCOMES:
Measurement of the Effective reproduction rate R in CAR according to the level of immunity (smallpox vaccine immunity or orthopoxvirus-related post disease immunity). | 36 months
  measurement of the level of population natural immunity and post vaccinal immunity to determine the Effective reproduction rate R and changes in R between 2000-2020 according to the evolution of immunity (smallpox vaccine immunity or orthopoxvirus-related post disease immunity).
measurement of the sensitivity and the specificity of the existing diagnostic tests and those developed within the framework of the project | 36 months
  sensitivity and specificity of the existing diagnostic tests and those developed within the framework of the project, as well as the reproducibility of measurements in relation to reference tests.
Identification and interpretation of genomic viral mutations from the viral sequences isolated from humans and animals in CAR for Phylogenetic and phylogeographic study of the monkeypox virus | 36 months
  identification and interpretation of mutations, search for the common ancestor.
Comparison of genetic proximities between different viral strains isolated in humans and animals in CAR and neighboring countries since 1980. | 36 months
  Comparison of genetic proximities
Identification of the characteristics associated with the environments in which human cases of monkeypox virus infection have occurred | 36 months
  ecosystems and their recent modifications, land use, associated climatic/meteorological elements in the tropical zone (CAR, Northern DRC...).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pasteur Bangui, Bangui, Central African Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Besombes C, Gonofio E, Konamna X, Selekon B, Grant R, Gessain A, Berthet N, Manuguerra JC, Fontanet A, Nakoune E. Intrafamily Transmission of Monkeypox Virus, Central African Republic, 2018. Emerg Infect Dis. 2019 Aug;25(8):1602-1604. doi: 10.3201/eid2508.190112. Epub 2019 Aug 17. PMID 31216261
- [Background] Berthet N, Descorps-Declere S, Besombes C, Curaudeau M, Nkili Meyong AA, Selekon B, Labouba I, Gonofio EC, Ouilibona RS, Simo Tchetgna HD, Feher M, Fontanet A, Kazanji M, Manuguerra JC, Hassanin A, Gessain A, Nakoune E. Genomic history of human monkey pox infections in the Central African Republic between 2001 and 2018. Sci Rep. 2021 Jun 22;11(1):13085. doi: 10.1038/s41598-021-92315-8. PMID 34158533
- See also: Institut Pasteur Afripox — https://research.pasteur.fr/fr/project/afripox/